CLINICAL TRIAL: NCT01837056
Title: Prevalence of Toxoplasma Gondii and Toxocara Canis Among Patients With Uveitis
Status: Completed | Type: Observational
Sponsor: National Institute of Health, Korea (Other Government)
Responsible Party: Principal Investigator, Lim, Su Jin, The retina staff, Nune Eye Hospital, Seoul, Korea
Other Study IDs: Nuneuveitis
Record Dates: First submitted 2013-04-12; First posted 2013-04-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Uveitis
Keywords: Toxoplasma gondii; Toxocara canis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Investigate the prevalence of Toxoplasma gondii and Toxocara canis in Uveitis

* serum antibody to T. gondii and T. canis
* PCR with peripheral blood for T. gondii and T. canis
* PCR with aqueous humor for T. gondii and T. canis
* Clinical manifestation of patient with uveitis

DETAILED DESCRIPTION:
Consecutive patients with uveitis are enrolled in Nune Eye Hospital.

Serum ELISA

* IgM,IgG antibody to Toxoplasma gondii
* IgG antibody to Toxocara canis

PCR

* PCR with serum and aqueous humor to Toxoplasma gondii
* PCR with serum and aqueous humor to Toxocara canis Clinical characteristics
* visual acuity
* intraocular pressure (IOP)
* location and degree of inflammation
* other fundus findings were recorded

questionnaire

* environment, occupation
* pet ownership, exposure to animal
* history of eating raw liver of animal, raw beef or any other raw flesh of animal.

ELIGIBILITY:
Inclusion Criteria:

* patients with uveitis

Exclusion Criteria:

* Patients with history of major ophthalmic surgery within 6 months
* antiviral, antifungal or antiparasitic therapy within 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patient with uveitis
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2011-01; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Number of patients with positive result for serum antibody to Toxoplasma gondii and Toxocara canis | at baseline
  proportion of patients with seropositive for Toxoplasma gondii and Toxocara canis among patients

SECONDARY OUTCOMES:
Number of patients with positive PCR with peripheral blood and aqueous humor to Toxoplasma gondii and Toxocara canis | at baseline
  Proportion of patient with positive PCR to Toxoplasma gondii and Toxocara canis

OTHER OUTCOMES:
location of inflammation and fundus finding | at baseline
  location of inflammation
  * anterior or posterior or panuveitis
  fundus finding
  * granuloma in macular or periphery retina
  * pigmentation
Demographic characteristics | at baseline
  * Gender
  * Residence
  * Pet ownership
  * Habit of eating uncooked meat

CONTACTS AND LOCATIONS:
Overall Officials: Su Jin Lim, MD, Principal Investigator — Nune Eye Hospital